CLINICAL TRIAL: NCT05448963
Title: A Pilot Study of Robot-assisted Nipple-sparing Mastectomy Followed by Immediate Breast Reconstruction Using da Vinci SP ® Single-port System
Brief Title: Pilot Study of Single-port Robot-assisted Nipple-sparing Mastectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Intuitive Surgical (Industry)
Responsible Party: Principal Investigator, KUO, WEN-LING, Director of Breast Cancer Center, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202101421A0
Record Dates: First submitted 2022-06-18; First posted 2022-07-08 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Nipple-sparing Mastectomy; Prophylactic Mastectomy; Breast Cancer; BRCA1 Mutation; BRCA2 Mutation
Keywords: robotic mastectomy; robot-assisted mastectomy; nipple-sparing mastectomy; axillary lymph node dissection; breast cancer surgery; breast reconstruction; prophylactic mastectomy; single-port systems
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: single arm surgical intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Robotic mastectomy (Experimental): Patients receive unilateral or bilateral robot-assisted nipple-sparing mastectomy with or without axillary lymph node dissection
  Interventions: Device: da Vinci SPⓇ Single-port System

INTERVENTIONS:
Device: da Vinci SPⓇ Single-port System — Nipple-sparing mastectomy with or without axillary lymph node dissection using da Vinci SP single-port system

SUMMARY:
Nipple-sparing mastectomy (NSM) is indicated for breast cancer requiring total mastectomy and without nipple involvement by cancer. Robot-assisted mastectomy enables removal of the whole breast tissue with well-preserved breast skin envelope through a single longitudinal incision in the anterior axillary line at the nipple areolar level. The next-generation robot, da Vinci SP system, is single-armed, equipped with multiple flexible instruments and camera, which is likely to improve the efficacy of robotic mastectomy. The investigator's scope of this study is to establish the feasibility and safety of SP-applied NSM through this single-armed pilot trial. Participants with breast cancer indicated for nipple-sparing mastectomy or candidates of prophylactic mastectomy carrying germline pathogenic or likely pathogenic BRCA1/2 mutations are recruited to receive SP-assisted unilateral or bilateral NSMs. Immediate breast reconstruction is followed according to the mode of the plastic surgeon's clinical decision. The primary endpoint is technical feasibility, and the secondary endpoint is safety and patient-reported outcome.

DETAILED DESCRIPTION:
About 49% of breast cancer surgery is managed by total mastectomy, and half of the patients undergo breast reconstruction. Nipple-sparing mastectomy (NSM) is indicated for breast cancer requiring total mastectomy and without nipple involvement by cancer. The local recurrence rate is not increased and the cosmetic result much improved. Robot-assisted mastectomy utilizes surgeon-controlled robotic arms with delicate, multi-jointed instruments and 3-dimentional high-definition camera in place of conventional instruments under bare eye vision. Through a single longitudinal incision in the anterior axillary line at the nipple areolar level, the lesion and the whole breast tissue can be totally removed with negative resection margins and well-preserved breast skin envelope. Breast reconstruction can be successfully performed through the same incision and results in a scarless front view. Currently, this surgery is effectively carried out with da Vinci Xi system. However, the small incision may result in the collision of robotic arms outside the torso and hence decreases the range of instrument motion. The next-generation robot, da Vinci SP system, is single-armed, equipped with multiple flexible instruments and camera, which are devoid of outside collision and allows work in a larger surgical field through the same small incision. The SP system reduces blind areas in the surgical field and the blockade of camera vision by the detached space-taking specimens, and, therefore, will hopefully reduce the surgical time. The investigator's scope of this study is to establish the feasibility and safety of SP-applied NSM through this single-armed pilot trial. The investigators recruit breast cancer women indicated for nipple-sparing mastectomy or candidates of prophylactic mastectomy carrying germline pathogenic or likely pathogenic BRCA1/2 mutations to receive SP-assisted unilateral or bilateral NSMs. Immediate breast reconstruction is followed according to the mode of the plastic surgeon's clinical decision. The primary endpoint is technical feasibility (conversion rate, surgical time), and the secondary endpoint is safety and patient-reported outcome.

ELIGIBILITY:
Inclusion Criteria:

* Women with unilateral or bilateral breast cancer, including invasive and noninvasive carcinoma, eligible for unilateral or bilateral nipple-sparing mastectomy (NSM), either for therapeutic or prophylactic purpose, followed by immediate breast reconstruction.

  1. Meet at least one of the following indications of NSM for breast cancer:

     1. Preoperative clinical tumor sizes less than 5 cm, with adequate tumor-skin distance of at least 3mm and above, and without nipple-areolar involvement in at least 1cm around the nipple by image
     2. Breast cancer up to stage IIIa (T3, N1-2) as the initial clinical stage showing adequate response to neoadjuvant therapy and meet criteria a.
     3. Germline pathogenic/likely pathogenic BRCA1 or 2 mutation carriers (actionable mutations including pathogenic and likely pathogenic mutations) with breast cancer diagnosis or requiring unilateral or bilateral prophylactic mastectomy as a risk reduction procedure
  2. Age equal to or above 20 years
  3. ECOG (Eastern Cooperative Oncology Group) performance score 0-1
  4. ASA anesthesia risk class 1~2, and with adequate organ functions
  5. Understanding of the method, benefit and risk and willing to receive immediate breast reconstruction

Exclusion Criteria:

1. Extensive breast skin or nipple involvement by cancer including 1) Paget's disease, 2) nipple discharge associated with malignancy, 3) image findings suggesting involvement of the nipple and subareolar tissues 4) inflammatory breast cancer or skin ulceration caused by cancer invasion
2. Stage III (up to T3, N1-2) breast cancer without response to neoadjuvant treatment
3. Previous radiotherapy on the surgical site of breast
4. Patients with severe systemic disease reaching ASA (American Society of Anesthesiologists) physical status classification equal or greater than 3
5. Patients with bleeding disorder or coagulopathy
6. Patients with BMI 35.0 or higher
7. Patients with habitual smoking
8. Pregnancy

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-30 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Surgical performance | Day 1
  Ability in percentage to complete nipple-sparing mastectomy with da Vinci SP system (no conversion to conventional laparoscopic, multiport da Vinci surgery or open surgery; addition of access port to complete the procedure would not be considered as conversion) in per protocol population

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Acute Complications | Day 1-Day 30
  Rate of incidence of surgery-related acute complications including hemorrhage, infection, skin ischemia, nipple ischemia, flap ischemia, and requirement for debridement or re-operation within 30 days
Incidence of Treatment-Emergent Mortality and Morbidity | Day 1-Day 30
  Morbidity and mortality rate resulting from surgery among per protocol population

OTHER OUTCOMES:
Blood loss | Day 1
  Blood loss in milliliters resulting from SP robotic mastectomy, and breast reconstruction respectively
Surgical time | Day 1
  Time in minutes consumed by robotic mastectomy and robotic operation: total surgical time, docking time, console operation time, mastectomy time, lymph node dissection time, reconstruction time
Body mass index | Day 0-1
  Patient weight and height to report BMI in kg/m^2
Specimen weight | Day 1
  Mastectomy specimen weight in miligrams
Mastectomy incision | Day 1
  Location and length in centimeters of robotic mastectomy incision
Oncological safety | Day 1-Day 30
  The ability to achieve margin-free resection for cancer cases: 1) Resection margin positive rate, 2) Nipple margin positive rate, 3)Nipple areolar complex excision rate (pre-planned, or based on nipple margin status, 4)Axillary surgery type (sentinel lymph node biopsy or axillary lymph node dissection)
Reconstructive surgery | Day 1-Day 2
  Type and status of concomitant breast reconstruction: 1) Type of reconstructive surgery (implant or autologous) 2) Impact reconstruction (if applicable): implant location, implant size/shape, brand/surface texture, or tissue expander location 3) Autologous reconstruction (if applicable): type of autologous tissue used, microsurgery detail, nipple neurotization detail
Drain output | Day 2-15
  Daily drain output in milliliters
Duration of admission | Day 0-60
  Total duration of admission in days for robotic mastectomy and immediate breast reconstruction
Long term complications | Day 90~
  Rate of complications resulting from robotic mastectomy and concomitant reconstruction more than 3 months after surgery
Patient-reported esthetic outcome | Day0, Day30, Day90, Day180, and Day360
  Serially evaluated patient-reported scores from Breast Q questionnaire
Patient-reported quality of life outcome for breast cancer cases | Day0, Day30, Day90, Day180, and Day360
  Serially evaluated patient-reported scores from EORTC-QLQ-C30 including functional and symptomatic scales comprising 30 items. The raw scores are linearly converted to a 0-100 scale, where higher function scores reﬂect more interfered function and higher symptom scores present a higher level of symptoms.
Patient-reported breast-specific quality of life outcome for breast cancer cases | Day0, Day30, Day90, Day180, and Day360
  Serially evaluated patient-reported scores from EORTC-QLQ-B23 including functional and symptomatic scales comprising 23 items. The raw scores are linearly converted to a 0-100 scale, where higher function scores reﬂect more interfered function and higher symptom scores present a higher level of symptoms.
Postoperative pain | Day2, Day4, Day6, Day8, Day15
  Serially evaluated intensity of pain by Numerical Rating Scale (Visual Analog Score) for pain, with scales ranging from 0-10. The intensity of pain increases with higher numerical scores (eg.,no pain(0), moderate pain (5), worst pain (10)).
Physician-evaluated outcomes | Picture taken on Day0, Day30, Day90, Day180, and Day360
  Questionnaires about post-reconstructive breast cosmesis evaluated by independent plastic surgeon through a Likert 5-point scale after reviewing pre-and post-operative pictures, where higher scale indicating higher cosmetic satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Ling Kuo, MD. PhD., Principal Investigator — Breast Cancer Center, Chang Gone Memorial Hospital , Linkou Medical Center
Locations (1):
- Chang Gung Memeorial Hospital, Linkou Medical Center, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD are to be shared upon request to the principle investigator. The content of data sharing depend on research relevance and cooperative detail.

REFERENCES:
- [Background] Sarfati B, Toesca A, Roulot A, Invento A. Transumbilical Single-port Robotically Assisted Nipple-sparing Mastectomy: A Cadaveric Study. Plast Reconstr Surg Glob Open. 2020 May 27;8(5):e2778. doi: 10.1097/GOX.0000000000002778. eCollection 2020 May. PMID 33133886
- [Background] Park HS, Lee J, Lee H, Lee K, Song SY, Toesca A. Development of Robotic Mastectomy Using a Single-Port Surgical Robot System. J Breast Cancer. 2020 Feb;23(1):107-112. doi: 10.4048/jbc.2020.23.e3. PMID 32140275
- [Background] Garcia-Etienne CA, Cody Iii HS 3rd, Disa JJ, Cordeiro P, Sacchini V. Nipple-sparing mastectomy: initial experience at the Memorial Sloan-Kettering Cancer Center and a comprehensive review of literature. Breast J. 2009 Jul-Aug;15(4):440-9. doi: 10.1111/j.1524-4741.2009.00758.x. Epub 2009 May 22. PMID 19496781
- [Background] Galimberti V, Vicini E, Corso G, Morigi C, Fontana S, Sacchini V, Veronesi P. Nipple-sparing and skin-sparing mastectomy: Review of aims, oncological safety and contraindications. Breast. 2017 Aug;34 Suppl 1(Suppl 1):S82-S84. doi: 10.1016/j.breast.2017.06.034. Epub 2017 Jun 30. PMID 28673535
- [Background] Shimo A, Tsugawa K, Tsuchiya S, Yoshie R, Tsuchiya K, Uejima T, Kojima Y, Shimo A, Hayami R, Nishikawa T, Yabuki Y, Kawamoto H, Sudo A, Fukuda M, Kanemaki Y, Maeda I. Oncologic outcomes and technical considerations of nipple-sparing mastectomies in breast cancer: experience of 425 cases from a single institution. Breast Cancer. 2016 Nov;23(6):851-860. doi: 10.1007/s12282-015-0651-6. Epub 2015 Oct 13. PMID 26464007
- [Background] Frey JD, Salibian AA, Levine JP, Karp NS, Choi M. Incision Choices in Nipple-Sparing Mastectomy: A Comparative Analysis of Outcomes and Evolution of a Clinical Algorithm. Plast Reconstr Surg. 2018 Dec;142(6):826e-835e. doi: 10.1097/PRS.0000000000004969. PMID 30204677
- [Background] Daar DA, Abdou SA, Rosario L, Rifkin WJ, Santos PJ, Wirth GA, Lane KT. Is There a Preferred Incision Location for Nipple-Sparing Mastectomy? A Systematic Review and Meta-Analysis. Plast Reconstr Surg. 2019 May;143(5):906e-919e. doi: 10.1097/PRS.0000000000005502. PMID 30789474
- [Background] Toesca A, Peradze N, Galimberti V, Manconi A, Intra M, Gentilini O, Sances D, Negri D, Veronesi G, Rietjens M, Zurrida S, Luini A, Veronesi U, Veronesi P. Robotic Nipple-sparing Mastectomy and Immediate Breast Reconstruction With Implant: First Report of Surgical Technique. Ann Surg. 2017 Aug;266(2):e28-e30. doi: 10.1097/SLA.0000000000001397. No abstract available. PMID 28692558
- [Background] Selber JC. Robotic Nipple-Sparing Mastectomy: The Next Step in the Evolution of Minimally Invasive Breast Surgery. Ann Surg Oncol. 2019 Jan;26(1):10-11. doi: 10.1245/s10434-018-6936-1. Epub 2018 Nov 12. No abstract available. PMID 30421063
- [Background] Toesca A, Peradze N, Manconi A, Galimberti V, Intra M, Colleoni M, Bonanni B, Curigliano G, Rietjens M, Viale G, Sacchini V, Veronesi P. Robotic nipple-sparing mastectomy for the treatment of breast cancer: Feasibility and safety study. Breast. 2017 Feb;31:51-56. doi: 10.1016/j.breast.2016.10.009. Epub 2016 Nov 2. PMID 27810700
- [Background] Lai HW, Wang CC, Lai YC, Chen CJ, Lin SL, Chen ST, Lin YJ, Chen DR, Kuo SJ. The learning curve of robotic nipple sparing mastectomy for breast cancer: An analysis of consecutive 39 procedures with cumulative sum plot. Eur J Surg Oncol. 2019 Feb;45(2):125-133. doi: 10.1016/j.ejso.2018.09.021. Epub 2018 Oct 17. PMID 30360987
- [Background] Lai HW, Lin SL, Chen ST, Kuok KM, Chen SL, Lin YL, Chen DR, Kuo SJ. Single-Axillary-Incision Endoscopic-Assisted Hybrid Technique for Nipple-Sparing Mastectomy: Technique, Preliminary Results, and Patient-Reported Cosmetic Outcome from Preliminary 50 Procedures. Ann Surg Oncol. 2018 May;25(5):1340-1349. doi: 10.1245/s10434-018-6383-z. Epub 2018 Feb 26. PMID 29484564
- [Background] Lai HW, Toesca A, Sarfati B, Park HS, Houvenaeghel G, Selber JC, Cheng FT, Kuo WL, Peradze N, Song SY, Mok CW. Consensus Statement on Robotic Mastectomy-Expert Panel From International Endoscopic and Robotic Breast Surgery Symposium (IERBS) 2019. Ann Surg. 2020 Jun;271(6):1005-1012. doi: 10.1097/SLA.0000000000003789. PMID 31977514
- [Background] Kuo WL, Huang JJ, Huang YT, Chueh LF, Lee JT, Tsai HP, Chen SC. Robot-assisted Mastectomy Followed by Immediate Autologous Microsurgical Free Flap Reconstruction: Techniques and Feasibility in Three Different Breast Cancer Surgical Scenarios. Clin Breast Cancer. 2020 Feb;20(1):e1-e8. doi: 10.1016/j.clbc.2019.06.018. Epub 2019 Sep 4. No abstract available. PMID 31780382
- [Background] Toesca A, Sangalli C, Maisonneuve P, Massari G, Girardi A, Baker JL, Lissidini G, Invento A, Farante G, Corso G, Rietjens M, Peradze N, Gottardi A, Magnoni F, Bottiglieri L, Lazzeroni M, Montagna E, Labo P, Orecchia R, Galimberti V, Intra M, Sacchini V, Veronesi P. A Randomized Trial of Robotic Mastectomy Versus Open Surgery in Women With Breast Cancer or BrCA Mutation. Ann Surg. 2022 Jul 1;276(1):11-19. doi: 10.1097/SLA.0000000000004969. Epub 2021 Jun 9. PMID 34597010
- [Background] Lemaine V, Hoskin TL, Farley DR, Grant CS, Boughey JC, Torstenson TA, Jacobson SR, Jakub JW, Degnim AC. Introducing the SKIN score: a validated scoring system to assess severity of mastectomy skin flap necrosis. Ann Surg Oncol. 2015 Sep;22(9):2925-32. doi: 10.1245/s10434-015-4409-3. Epub 2015 Jan 30. PMID 25634782
- [Background] Joo OY, Song SY, Park HS, Roh TS. Single-port robot-assisted prosthetic breast reconstruction with the da Vinci SP Surgical System: first clinical report. Arch Plast Surg. 2021 Mar;48(2):194-198. doi: 10.5999/aps.2020.01557. Epub 2021 Mar 15. PMID 33765738
- [Background] Lee J, Park HS, Lee H, Lee K, Han DH, Lee DW. Axillary lymph node dissection using a robotic surgical system: Initial experience. J Surg Oncol. 2020 Nov;122(6):1252-1256. doi: 10.1002/jso.26141. Epub 2020 Aug 11. No abstract available. PMID 32783194
- [Background] Huang JJ, Chuang EY, Cheong DC, Kim BS, Chang FC, Kuo WL. Robotic-assisted nipple-sparing mastectomy followed by immediate microsurgical free flap reconstruction: Feasibility and aesthetic results - Case series. Int J Surg. 2021 Nov;95:106143. doi: 10.1016/j.ijsu.2021.106143. Epub 2021 Oct 16. PMID 34666195